CLINICAL TRIAL: NCT00690196
Title: Tai Chi Effects on Chronic Insomnia in Breast Cancer Survivors: Immune Mechanism
Brief Title: Tai Chi Effects on Chronic Insomnia in Breast Cancer Survivors: Immune Mechanisms
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: National Center for Research Resources (NCRR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 11-000625; M01RR000865 (NIH); R01 CA119 159 (Other Grant/Funding Number: NCI)
Record Dates: First submitted 2008-03-10; First posted 2008-06-04 (Estimated); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Sleep Disorders; Sleep Initiation and Maintenance Disorders; Dyssomnias; Mental Disorders; Nervous System Diseases
MeSH Terms: conditions — Sleep Wake Disorders; Sleep Initiation and Maintenance Disorders; Dyssomnias; Mental Disorders; Nervous System Diseases | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Tai Chi Chih
  Interventions: Behavioral: Tai Chi Chih
- 2 (Active Comparator): Cognitive Behavioral Therapy
  Interventions: Behavioral: Cognitive Behavioral Therapy

INTERVENTIONS:
Behavioral: Tai Chi Chih — Tai Chi Chih (TCC) employs "meditation through movement" as a means of helping breast cancer survivors cope with fatigue, perceived physical limitations, and negative emotional states which are commonly associated with insomnia. In groups of 7-8, subjects will learn to perform 20 movements under the guidance of expert TCC teacher (K. Hollister, certified instructor) who will oversee treatment sessions throughout the 12 week treatment, consistent with our preliminary studies (9). Sessions will be taught over 120 minutes with 90 minutes of active TCC, 20 minutes of warm-up (e.g., stretching, breathing),10 minutes of cool down. Sessions will be mainly given in the late afternoon at 16:00 h. Thus, the TCC will be given once a week per week for a total of 120 minutes, similar in total time allocation with Cognitive Behavioral Therapy. The final week of treatment will include the development of a TCC adherence plan to ensure continuity of practice and skill maintenance during follow-up.
  Other Names: TCC
  Arms: 1
Behavioral: Cognitive Behavioral Therapy — Cognitive Behavioral Therapy (CBT) for insomnia will be supervised by a Ph.D. level psychologist, with specialty training in behavior therapy and behavioral medicine. The CBT sessions will be held once a week for 120 minutes (each session) over the 12-week treatment period, identical to the time schedule which was to be used for health education. Treatment will be given in small groups of 7-8 subjects. The content of the intervention will be organized around a series of modules that will be presented to patients in manualized form. For each session, the CBT treatment manual will outline objectives, patient skills, and treatment activities. Therapists will direct role-playing and other skill-development exercises that will be designed to increase patients' self-efficacy in managing their insomnia. Homework assignments will be planned weekly to ensure practice and skill application.
  Other Names: CBT
  Arms: 2

SUMMARY:
Breast Cancer is the most common cancer in women. After completion of successful therapy, may behavioral symptoms persist with over 20% of breast cancer survivors reporting chronic insomnia of greater than 6 months duration that fulfils clinical diagnostic criteria with associated functional limitations, decreased quality of life, and possible effects on long-term survival. Behavioral interventions are highly efficacious in the treatment of insomnia and preferred over hypnotic medication when insomnia is chronic. However, insomnia studies conducted in cancer are scarce. The proposed research builds upon program of study that has examined the efficacy of mind-body intervention, Tai Chi Chih (TCC), on health outcomes including sleep impairments. Preliminary studies show that TTC, a slow moving meditation, contributes to improvement in subjective sleep quality, sleep amounts and sleep efficiency. The investigators have further found that sleep, fatigue and proinflammatory cytokine activity are reciprocally related and that TCC decreases the mechanism through TCC carries its effects on sleep outcomes.

DETAILED DESCRIPTION:
This investigation is a randomized controlled trial that will evaluate the effects of cognitive-behavioral therapy (CBT) and Tai Chi Chih (TCC) on objective and subjective measures of sleep, on mood and fatigue, on health functioning and on two biological parameters, sympathovagal tone and proinflammatory cytokine activity in older adults with insomnia. One hundred breast cancer survivors will be randomly assigned to CBT, or TCC. Patients will be assessed at pre-treatment, during midtreatment, post-treatment, 3-month follow-up and 12-month follow-up. At all 5 assessment periods, indices of sleep quality as measured by sleep diaries and clinical ratings will be obtained along with measures of mood, health functioning, proinflammatory cytokine activity and heart rate variability (HRV). The pre-treatment and post-treatment assessment periods will also include all-night polysomnography along with nocturnal sampling of proinflammatory cytokine activity and HRV tone. Hence, polysomnographic measures of sleep which are coupled with nocturnal measures of cytokines by serial blood sampling will occur at the baseline assessment and again at the post-treatment assessment. During midtreatment and at 3 month follow-up and 12 month follow-up, we will obtain questionnaire ratings of sleep quality along with a single morning sample of cytokine levels.

ELIGIBILITY:
Inclusion Criteria:

* 100 postmen women between the ages of 30 - 70 years who were originally diagnosed with early, resectable breast cancer (Stage 0, I, or II, III), have completed treatment with surgery, radiation, and/or chemotherapy, and show no evidence of cancer recurrence or new primary tumor.
* Difficulty sleeping for a minimum of 3 nights per week
* Insomnia duration at least 6 months
* Complaint of at least 1 negative effect during waking hours (e.g. fatigue, impaired functioning, mood disturbances) attributed to insomnia
* Habitual sleep-wake schedule reporting "lights-out" between 9:00 PM-midnight
* Accessible geographically

Exclusion Criteria:

* Evidence that insomnia is directly related to a medical disorder (e.g., hyperthyroidism) or effects of a medication that affects sleep structure and/or immune functioning
* Presence of sleep apnea (apnea-hypopnea index >15) or periodic limb movements during sleep (myoclonic index with arousal >15) as assessed by PSG;
* Presence of another sleep disorder (e.g., Advanced or Delay Sleep Phase Syndrome)
* Current or History of another major psychiatric disorder
* Cognitive impairment as suggested by a score lower than 23 on the Mini-Mental State examination;
* Smokers will also be excluded because of potential confounding effects on markers of inflammation;
* Body mass index that is greater than 35 kg/m2, obesity is associated with excessive levels of inflammatory markers
* Unable to commit to intervention schedule.

Ages: 30 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2008-03; Primary Completion 2026-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Changes in insomnia symptoms as measured by subjective report and objective polysomnography; Changes in daytime impairment secondary to insomnia; Changes in fatigue, depression and mood, and health function | 5 years

SECONDARY OUTCOMES:
Overall Health and Well-being | 5 years
  Changes in sympathovagal function and energy balance; Changes in measures of interpersonal resilience and social functioning; physical activity; cognitive function; mental health
Allostatic Load | 5 years
  Measure of metabolic and allostatic load will be assesed with clinical laboratory tests.
Inflammatory Markers | 5 years
  Changes in measure of proinflammatory cytokines activity;

CONTACTS AND LOCATIONS:
Overall Officials: Michael Irwin, MD, Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA Cousins Center for Psychoneuroimmunology, Los Angeles, California, United States

REFERENCES:
- [Background] Irwin MR, Olmstead R, Oxman MN. Augmenting immune responses to varicella zoster virus in older adults: a randomized, controlled trial of Tai Chi. J Am Geriatr Soc. 2007 Apr;55(4):511-7. doi: 10.1111/j.1532-5415.2007.01109.x. PMID 17397428
- [Background] Bower JE, Ganz PA, Aziz N, Olmstead R, Irwin MR, Cole SW. Inflammatory responses to psychological stress in fatigued breast cancer survivors: relationship to glucocorticoids. Brain Behav Immun. 2007 Mar;21(3):251-8. doi: 10.1016/j.bbi.2006.08.001. Epub 2006 Sep 27. PMID 17008048
- [Background] Motivala SJ, Sarfatti A, Olmos L, Irwin MR. Inflammatory markers and sleep disturbance in major depression. Psychosom Med. 2005 Mar-Apr;67(2):187-94. doi: 10.1097/01.psy.0000149259.72488.09. PMID 15784782
- [Background] Irwin MR, Pike JL, Cole JC, Oxman MN. Effects of a behavioral intervention, Tai Chi Chih, on varicella-zoster virus specific immunity and health functioning in older adults. Psychosom Med. 2003 Sep-Oct;65(5):824-30. doi: 10.1097/01.psy.0000088591.86103.8f. PMID 14508027
- [Derived] Cai Z, Tang Y, Liu C, Li H, Zhao G, Zhao Z, Zhang B. Cognitive behavioural therapy for insomnia in people with cancer. Cochrane Database Syst Rev. 2025 Oct 31;10(10):CD015176. doi: 10.1002/14651858.CD015176.pub2. PMID 41170811